CLINICAL TRIAL: NCT01521039
Title: Assessment of MicroRNA Expression in Acute Graft-versus-Host Disease
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Hannah Choe, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-11002
Record Dates: First submitted 2012-01-23; First posted 2012-01-30 (Estimated); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Graft-versus-Host Disease; Allogeneic Stem Cell Transplant
Keywords: aGVHD; Acute Graft-versus-Host Disease; allogeneic stem cell transplantation; Hematopoietic stem cell transplantation; MicroRNA Expression
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Allogeneic SCT recipients: Patients who are receiving allogeneic stem cell transplantation at the Ohio State University are eligible and will be consented for the study.
  Interventions: Procedure: Blood samples

INTERVENTIONS:
Procedure: Blood samples — 2-3 tablespoons of blood weekly for the first 100 days (about 14 weeks) following allogeneic transplant. In addition a blood sample will be obtained before starting the chemotherapy or radiation regimen for the transplant, in the day of the transplant and if your doctor suspects that you have acute graft-versus-host disease.
  Other Names: peripheral blood; whole blood

SUMMARY:
Assessment of MicroRNA Expression in Acute Graft-versus-Host Disease (GVHD).

DETAILED DESCRIPTION:
The purpose of this study is to examine whether the expression levels of a novel class of molecules, called microRNAs, are associated with acute graft-versus-host disease frequency and severity. Acute graft-versus-host disease is a Acute GVHD is a medical condition that can become very serious. It happens when the donor cells attack and damage your tissues after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving allogeneic stem cell transplantation at the Ohio State University Blood and Marrow Transplantation program are eligible and will be consented for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are receiving allogeneic stem cell transplantation at the Ohio State University are eligible and will be consented for the study.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2012-02-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Measure miR-155 expression levels over time in the serum from patients receiving allogeneic stem cell transplant, and evaluate if miR-155 expression can predict development of aGVHD (Acute Graft-versus-Host Disease) | up to 14 weeks

SECONDARY OUTCOMES:
Compare miR-155 expression at the time of clinical suspicion of aGVHD in allogeneic recipients with aGVHD diagnosis with matched allogeneic recipients without aGVHD. | up to 14 weeks
Correlate miR-155 expression at the time of clinical suspicion of aGVHD in allogeneic recipients with the severity of aGVHD. | up to 15 weeks
Perform serum global microRNA analysis in allogeneic recipients at the time of clinical suspicion of aGVHD to identify other miRNAs that are associated with aGVHD diagnosis and severity. | up to 15 weeks
Collect and store serum/plasma and mononuclear cells from patients receiving allogeneic blood and marrow stem cell transplantation. | up to 14 weeks
  Perform the following: a) validation of the miRNA expression profiling signatures; b) correlation of miRNA expression among serum, plasma and mononuclear cells; and c) correlation of relevant miRNA targets or regulators expression (at the RNA or protein level) with miR-155 and other miRNAs expression identified in the aGVHD miRNA signatures.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Choe, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu